CLINICAL TRIAL: NCT06210659
Title: The The Effect of Planned Behavior Theory-Based Education Program Applied to University Students With Primary Dysmenorrhea on Physical Activity Behavior and the Level of Affected by Dysmenorrhea
Brief Title: The The Effect of Planned Behavior Theory-Based Education on Physical Activity and Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Aycin Cifci, PHD STUDENT, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AnkaraU-HEM-RK-01
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Dysmenorrhea Primary
Keywords: Dysmenorrhea; Theory of Planned Behavior; Physical Activity; Pain
MeSH Terms: conditions — Dysmenorrhea; Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: 2 groups; intervention and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Theory of Planned Behavior Based Training Program will be implemented. The training program will consist of 4 sessions. Students will be monitored for 3 menstrual cycles. Starting from the end of the first menstrual period after completion of the training session, students will be asked to record their daily step count using a pedometer. In each menstrual period, the average of the students' monthly step count and average menstrual pain score will be evaluated. After the training sessions are completed, students will be given an end-of-menstrual motivational interview for 3 menstrual cycles.
  Interventions: Behavioral: Theory of Planned Behavior Based Training Program
- Control group (No Intervention): Students will be required to record their daily step count using a pedometer. Students will be monitored for 3 menstrual cycles. In each menstrual period, the average of the students' monthly step count and average menstrual pain score will be evaluated.

INTERVENTIONS:
Behavioral: Theory of Planned Behavior Based Training Program — Theory of Planned Behavior Based Training Program will be implemented. The training program will consist of 4 sessions. First session; It will consist of the definition, symptoms and treatment approaches of primary dysmenorrhea. Content of the second session; It will consist of lifestyle interventions in dysmenorrhea. Content of the third session; It will consist of the importance of physical activity in primary dysmenorrhea. The fourth session consists of a group walk.
  Students will be monitored for 3 menstrual cycles. Starting from the end of the first menstrual period after completion of the training session, students will be asked to record their daily step count using a pedometer. In each menstrual period, the average of the students' monthly step count and average menstrual pain score will be evaluated. After the training sessions are completed, students will be given an end-of-menstrual motivational interview for 3 menstrual cycles.
  Arms: Intervention group

SUMMARY:
The aim of the study is to examine the effect of the planned behavior theory-based education program applied to university students with primary dysmenorrhea on physical activity behavior and dysmenorrhea's impact.

DETAILED DESCRIPTION:
The study was planned to be conducted as a randomized controlled experimental study in the pre-test-post-test order.

The research was planned to be conducted at Bitlis Eren University. The population of the research consists of first year students studying at the Faculty of Arts and Sciences, Faculty of Fine Arts, Faculty of Economics and Administrative Sciences, Faculty of Islamic Sciences, Faculty of Engineering and Architecture, who are studying at Bitlis Eren University in the 2023-2024 academic year.

The sample of the research will consist of 54 students who meet the inclusion criteria and agree to participate in the research. Considering the possible losses that may occur during the research process, a total of 68 students are planned to be accepted.

The research data were collected with; "Inclusion Criteria Questionnaire", "Exhibitor Introduction Form", "Visual Pain Scale", "Physical Activity Scale", "Dysmenorrhea Impact Scale Short Form", "The Self-Effıcacy Scale" and "Daily Step Tracking Form".

In the research, Planned Behavior Theory Based Training Program consisting of 4 sessions will be applied to the intervention group, and information will be given to the control group about the process of the research and the data collection forms to be used. Students in both groups will have 3 menstrual cycles after the education.

In the study, it is planned to use descriptive statistics (number, percentage, mean and standard deviation) in the analysis of quantitative data, t test and Mann Whitney U test in the comparison of paired groups, Mcnemar test in the comparison of two groups, analysis of variance in the comparison of multiple groups, and Pearson and Spearman correlation analysis in relational inferences.

ELIGIBILITY:
Inclusion Criteria:

* Last menstrual pain is 5 points or more out of 10 on the Visual Pain Scale (moderate/severe/unbearable pain),
* Being 18 years or older,
* Reading and writing Turkish,
* Receiving education at undergraduate level,
* Being a first year student,
* Being nulliparous (never giving birth) and never having had a pregnancy,
* Having a regular menstrual cycle (every 21-35 days, lasting 3-8 days and without complaints of intermittent bleeding) for the last 6 months,
* Being inactive or minimally active according to the International Physical Activity Survey,
* Being diagnosed with primary dysmenorrhea by the physician,
* Agreeing to participate in the study.

Exclusion Criteria:

* Receiving education at the health vocational high school level,
* Last menstrual pain is 4 points or less out of 10 on the Visual Pain Scale,
* Having any gynecological diagnosis (endometriosis, ovarian cyst, myoma, polyp, etc.),
* Having undergone a gynecological operation (hysterectomy, myomectomy, etc.),
* Being on hormonal drug therapy,
* Having an orthopedic disability (congenital limb deficiencies, congenital hip dislocation, scoliosis, meningomyolocele, cerebral palsy, etc.), visual disability (vision loss, peripheral retinopathy, hemianopia, night blindness, etc.) and hearing disability that would prevent physical activity,
* Having acute or severe pain that increases with movement,
* Having a known systemic and chronic disease (diabetes, heart disease, vascular diseases, circulatory disorders, varicose veins, blood diseases, etc.),
* Having any psychiatric diagnosis (depression, anxiety disorder, etc.)
* Not agreeing to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Due to women experiencing primary dysmenorrhea.
Enrollment: 68 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 4 MONTHS
  "0" IS DEFINED AS NO PAIN, "10" IS DEFINED AS VERY SEVERE PAIN. AS THE VALUE INCREASES, THE SEVERITY OF PAIN INCREASES.

SECONDARY OUTCOMES:
Dysmenorrhea Impact Scale-Short Form | 4 MONTHS
  It consists of 13 items. The scale is five-point Likert type. As the score obtained from the scale increases, the level of individuals being affected by dysmenorrhea also increases.
Physical Activity Scale | 4 MONTHS
  It was developed based on the "Theory of Planned Behavior". It consists of 30 items. As the total score average obtained from the physical activity scale increases, knowledge, behavior and status towards physical activity increase positively.
The Self-Effıcacy Scale | 4 MONTHS
  It consists of 23 items. Five-point Likert type scale. A high total score indicates that the general self-efficacy-sufficiency perception is high.
Daily Step Tracking | 4 MONTHS
  The daily step count will be recorded with the pedometer. The monthly average number of steps will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Demirtas, PhD, Principal Investigator — Ankara University
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No